CLINICAL TRIAL: NCT00484965
Title: Erythrocyte-Mediated Drug Delivery for the Prevention of Restenosis After Coronary Artery Stent Implantation:TROY-Study
Brief Title: Erythrocyte-Mediated Drug Delivery for the Prevention of Stent Restenosis
Acronym: TROY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: University of Milan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 72/06
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Atherosclerosis; Acute-Phase Reaction
Keywords: Coronary stent; Inflammation; Atherosclerosis; Immunosuppressive
MeSH Terms: conditions — Atherosclerosis; Acute-Phase Reaction; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Coronary stenting

SUMMARY:
The purpose of this study is to determine whether erythrocyte mediated dexamethasone delivery reduces circulating inflammatory markers after coronary stent implantation and improves clinical and angiographic outcomes.

DETAILED DESCRIPTION:
In stent restenosis is still an unsolved problem. We know that principally in stent restenosis depends on myointimal proliferation, a biological process in which inflammatory mechanisms play a central role. We have previously demonstrated that immunosuppressive therapy with prednisone administered for 45 days after the stenting procedure reduced the incidence of restenosis at six months and clinical events at 12 months in high risk patients, with persistent higher C reactive protein levels after stenting implantation. But this therapy needs a high dosage glucocorticoids, and this is a contraindication in some subset of patients i.e. diabetics.

Recently a new method for the encapsulation of drugs into human autologous erythrocytes using an apparatus and a disposable kit has been developed. It's well known that blood erythrocytes change their membrane properties when in contact with suspensions of different osmotic values. So we developed a method to modify erythrocytes membrane properties so that they became porous and be able to absorb and then release some specific molecules. Experimental studies demonstrated that non diffusible pro-drug 21-phosphate dexamethasone can be loaded in human blood erythrocytes and then slowly dephosphorylated to the corresponding diffusible molecule to be released in human plasma. Once in-vivo due to the presence of the hydrophilic phosphate group, Dex 21-P encapsulated into RBCs cannot diffuse through RBC membrane until it is slowly dephosphorylated to the corresponding active corticosteroid by erythrocytes resident enzymes. The novelty and the advantages of this procedure are that the red blood cells act as a slow and constant drug delivery system so that, during the 30 days after the administration, there is always a low level of corticosteroid in plasma. When these erythrocytes are reinfused in the donor, they release in a continuous way a low and constant level of drug. This procedure has yet been used in some chronic inflammatory disease (i.e. bowel disease) in more than 1600 patients, with significant clinical improvement. The main objective of the study is 1) to evaluate if autologous erythrocytes modified as bioreceptor may be used to release glucocorticoids in blood circulation and 2) to reduce acute inflammatory proteins after coronary stent implantation with clinical and angiographic outcomes improvement. For this purpose 100 patients undergoing coronary artery stent implantation will be prospectively randomized in two groups:

1. group A: bare metal stent implantation and treatment by 50 ml of autologous erythrocytes charged with dexamethasone 21-P
2. group B: bare metal stent implantation and treatment by 50 ml of autologous erythrocytes not charged with dexamethasone 21-P The results of two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* coronary disease
* written informed consent
* coronary stenosis
* CRP baseline levels < 0,5 mg/dl

Exclusion Criteria:

* acute myocardial infarction
* coronary bypass grafting restenosis
* vessels diameter < 2,5 mm
* corticosteroids contraindications
* corticosteroids therapy 30 days before
* active infective disease
* connective disease
* pregnancy
* cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-07; Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Determine whether erythrocyte mediated dexamethasone delivery reduces circulating inflammatory markers after coronary stent implantation and improves reduction of acute phase reaction proteins | one year

SECONDARY OUTCOMES:
Reduction of myointimal proliferation and restenosis after stenting implantation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Versaci, MD, FACC, Principal Investigator — Tor Vergata University, Rome; Francesco Versaci, MD, FACC, Study Director — Tor Vergata University, Rome; Luigi Chiariello, MD, FACC, Study Chair — Tor Vergata University, Rome
Locations (1):
- Policlinico Tor Vergata, Rome, Italy

REFERENCES:
- [Background] Versaci F, Gaspardone A, Tomai F, Ribichini F, Russo P, Proietti I, Ghini AS, Ferrero V, Chiariello L, Gioffre PA, Romeo F, Crea F; Immunosuppressive Therapy for the Prevention of Restenosis after Coronary Artery Stent Implantation Study. Immunosuppressive Therapy for the Prevention of Restenosis after Coronary Artery Stent Implantation (IMPRESS Study). J Am Coll Cardiol. 2002 Dec 4;40(11):1935-42. doi: 10.1016/s0735-1097(02)02562-7. PMID 12475452